CLINICAL TRIAL: NCT02766114
Title: Carpal Tunnel Release Through Mini Transverse Approach
Acronym: CTRMTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Issa, Abdulhamid Sayed, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sayed Issa's Approach; NCT02726165 (obsolete NCT alias); NCT02766413 (obsolete NCT alias)
Record Dates: First submitted 2016-05-04; First posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Carpal Tunnel Syndrome; Carpal Tunnel Release; Carpal Tunnel Surgery; Carpal Tunnel Transverse Approach; CTS
Keywords: CTS; Carpal tunnel syndrome; Carpal tunnel release; Mini incision of carpal tunnel release; Cosmetic surgery of carpal tunnel syndrome; endoscopic carpal tunnel surgery; Carpal Tunnel Release Through Mini Transverse Approach; Dr. Sayed Issa's Approach; CTRMTA; OCTR; ECTR; Open Carpal Tunnel Release; Endoscopic Carpal Tunnel Release; Syria; Cosmetic; Safety; Rehabilitation,; Complications; Surgery; Satisfaction
MeSH Terms: conditions — Carpal Tunnel Syndrome; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Issa1 (Experimental): After local anesthesia, through transverse approach on the middle of dorsal wrist crease the incision is made for 1.5 cm length, then the subcutaneous fat is dissected, soon we see the the palmaris longus tendon or its connection with the carpal ligament , take the ulnar side of the palmaris longus tendon and cut the carpal ligament axillary by scalpel, not going deep with the scalpel to avoid medial nerve injury, soon we see the nerve, we use the scissors to cut the proximal part then the distal part of the carpal ligament by enclosing it between the blades of the scissors, now the full released carpal tunnel most be observed, and one stitch is enough, in this operation most be an assistant exist.
  Interventions: Procedure: Carpal tunnel release through Mini Transverse Approach

INTERVENTIONS:
Procedure: Carpal tunnel release through Mini Transverse Approach — Carpal tunnel release through a transverse cosmetic small incision over the distal wrist crease.

SUMMARY:
Carpal tunnel release through dorsal wrist crease Mini Transverse incision, about 1.5 cm length.

DETAILED DESCRIPTION:
Carpal tunnel release through a small approach on the distal wrist crease, it is about 1.5 cm, the benefits of this technique is less surgical traumatic and more tender, it takes less time for rehabilitation, so the patient can work next day of operation, and it has very cosmetic and gentle scar in results and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with Carpal Tunnel Syndrome refractory to conservative treatment
* Participant cooperation sufficient to operate under local anesthesia

Exclusion Criteria:

* Un controlled diabetes mellitus type 1 and 2
* Patients with non controlled Vascular hypertension
* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization
* Patients with history of Carpal Tunnel release surgery failure

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with post surgical trauma | Up to eight weeks

SECONDARY OUTCOMES:
Duration of rehabilitation period | Up to three weeks
Proportion of patients with cosmetic scar | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Sayed Issa's Clinic, Aleppo, Syria

IPD SHARING:
Plan to Share IPD: Yes